CLINICAL TRIAL: NCT02856724
Title: Early Amniotomy After Vaginal Prostaglandin E2 for Induction of Labor at Term: a Randomized Clinical Trial
Acronym: PGE2
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Ahmet Eser, medical doctor, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 145
Record Dates: First submitted 2016-08-02; First posted 2016-08-05 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Early Amniotomy, Unfavorable Cervix
MeSH Terms: interventions — Dinoprostone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early amniotomy and PGE2 (Experimental): 10 mg PGE2 vaginal ovul(Propess) Early amniotomy will be done in the early active phase of labor for early amniotomy group ( half of participants) when the cervix will be dilated 3 cm using the amniotomy hook.
  Interventions: Drug: PGE2
- PGE2 (Active Comparator): 10 mg PGE2 vaginal ovul(Propess)
  Interventions: Drug: PGE2

INTERVENTIONS:
Drug: PGE2 — 10 mg PGE2 vaginal ovul(Propess)
  Other Names: dinoprostone

SUMMARY:
This study evaluates the effectiveness and safety of early amniotomy after vaginal prostaglandin E2 for induction of labor at term. Early amniotomy will be done in the early active phase of labor for early amniotomy group ( half of participants) when the cervix will dilated 3 cm using the amniotomy hook. Amniotomy will not be done for control group(other half of participants) until the membranes rupture spontaneously.

DETAILED DESCRIPTION:
During induction of labour, amniotomy (defined as artificial rupture of fetal membranes) is commonly used in combination with induction of labor. However, there is a lack of data on both effectiveness and ideal timing of this procedure. Yet for patients with an unfavorable cervix, a sharply ripening agent may be considered. As is well known to all,prostaglandin works efficiently in cervical ripening and labor induction. So dinoprostone surely performs quite well in promoting cervical ripening and labor induction since its main component is prostaglandin E2 (PGE2).

ELIGIBILITY:
Inclusion criteria

1. singleton pregnancy,
2. gestational age ≥34 weeks,
3. intact membranes,
4. cephalic presentation,
5. bishop score ≤5,
6. had obstetrical indications for induction of labor,
7. had less than three uterine contractions in every 10 minutes.

Exclusion Criteria:

1. Patients who have contraindications for vaginal delivery,
2. previous uterine surgery,
3. fetal malpresentation,
4. multifetal pregnancy,
5. more than three contractions in 10 minutes,
6. contraindications to prostaglandins,
7. a category II or III fetal heart rate pattern,
8. anomalous fetus,
9. fetal demise
10. women with immediate delivery indications -

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2016-08; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
induction-to- delivery time | delivery (the length of time between the beginning of induction and the end of labor)

SECONDARY OUTCOMES:
mode of labor (vaginal or C-section) | delivery
successful induction | vaginal delivery within 24 h from the beginning of induction

CONTACTS AND LOCATIONS:
Overall Officials: evrim bostanci ergen, M.D., Study Director — Zeynep Kamil Maternity and Children's Training and Research Hospital, Department of Obstetrics and Gynecology, Istanbul, Turkey
Locations (1):
- Zeynep Kamil Woman and Child Diseases Education and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Ozkan S, Caliskan E, Doger E, Yucesoy I, Ozeren S, Vural B. Comparative efficacy and safety of vaginal misoprostol versus dinoprostone vaginal insert in labor induction at term: a randomized trial. Arch Gynecol Obstet. 2009 Jul;280(1):19-24. doi: 10.1007/s00404-008-0843-9. Epub 2008 Nov 26. PMID 19034471
- [Background] Wei S, Wo BL, Qi HP, Xu H, Luo ZC, Roy C, Fraser WD. Early amniotomy and early oxytocin for prevention of, or therapy for, delay in first stage spontaneous labour compared with routine care. Cochrane Database Syst Rev. 2013 Aug 7;2013(8):CD006794. doi: 10.1002/14651858.CD006794.pub4. PMID 23926074
- [Result] Makarem MH, Zahran KM, Abdellah MS, Karen MA. Early amniotomy after vaginal misoprostol for induction of labor: a randomized clinical trial. Arch Gynecol Obstet. 2013 Aug;288(2):261-5. doi: 10.1007/s00404-013-2747-6. Epub 2013 Feb 21. PMID 23430026
- See also: Related Info — http://nih.gov